CLINICAL TRIAL: NCT03685565
Title: Cosmetic Outcomes of Simple Facial Lacerations Repaired With Dermabond Compared With Dermabond With Underlying Steristrips: A Randomized Controlled Trial
Brief Title: Facial Lacerations Repaired With Dermabond Compared With Dermabond With Underlying Steristrips in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Erin D Munns, Fellow Physician, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-05-0081
Record Dates: First submitted 2018-09-17; First posted 2018-09-26 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Facial Laceration
Keywords: facial laceration; pediatric; dermabond; skin glue; steristrips; skin adhesive; scar; cosmesis
MeSH Terms: conditions — Cicatrix | interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Intervention Model Description: Experimental group: Dermabond with underlying steristrips. Control group: Dermabond alone
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dermabond with underlying steristrips (Experimental)
  Interventions: Procedure: Dermabond and steristrips
- Dermabond (Active Comparator)
  Interventions: Procedure: Dermabond

INTERVENTIONS:
Procedure: Dermabond and steristrips — Laceration repaired with Dermabond with underlying steristrips
  Arms: Dermabond with underlying steristrips
Procedure: Dermabond — Laceration repaired with Dermabond
  Arms: Dermabond

SUMMARY:
The purpose of the study is to compare cosmetic outcomes of simple facial lacerations in children repaired with Dermabond (skin glue) compared with Dermabond (skin glue) with underlying steristrips (skin adhesive strips).

ELIGIBILITY:
Inclusion Criteria:

* Age ≤17 years old
* Presents with simple, linear facial laceration requiring repair
* English or Spanish speaking parents or guardians

Exclusion Criteria:

* Laceration to lips, nose, ear, eyelids, eyebrows
* Laceration requiring multi-layer closure
* Laceration requiring sub-specialty care
* Laceration that has previously been repaired
* Animal/human bites
* Lacerations >5cm in length
* Allergy to adhesive

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Cosmesis | 2 months after repair
  cosmetic scar outcome; photo will be taken of scar at 2 months and graded using a visual analog scale (VAS) by blinded reviewers. The VAS is a 0-100mm standardized scale where 0mm represents the "worst scar" and 100mm represents the "best scar" and reviewers will place a marking along the line of where they feel the scar belongs.

SECONDARY OUTCOMES:
Time to repair laceration | Day 0 (physician will complete just after the repair)
  A stopwatch will be used to time how long it takes the physician to repair the wound
Ease of repair of laceration | Day 0 (physician will complete just after the repair)
  Physicians will complete a VAS (visual analog scale) on how easy the laceration was to repair. The VAS is a 0-100mm scale where 0 will represent "very easy" and 100mm will represent "very difficult" to repair and the physician will mark along the scale.
Type of analgesia & sedation required | Day 0 (physician will complete just after the repair)
  Physician will write down what types of analgesia they used and whether or not sedation was used after the repair is complete
Wound dehiscence | 1 week
  Families will get a phone call at 1 week to discuss if this has occurred. The electronic medical record will also be reviewed.
Wound infection | 1 week
  Families will get a phone call at 1 week to discuss if this has occurred. The electronic medical record will also be reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Munns, MD, Principal Investigator — University of Texas at Austin
Locations (1):
- Dell Children's Hospital, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munns E, Kienstra AJ, Combs PD, Gabriele G, Wilkinson M. Cosmetic Outcomes of Simple Pediatric Facial Lacerations Repaired With Skin Adhesive Compared With Skin Adhesive With Underlying Adhesive Strips: A Randomized Controlled Trial. Pediatr Emerg Care. 2022 Oct 1;38(10):477-480. doi: 10.1097/PEC.0000000000002837. Epub 2022 Aug 26. PMID 36018733